CLINICAL TRIAL: NCT01379092
Title: An Evaluation of a Self-contained Direct Digital Radiography System for Breast Specimen Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Levine, Gary M. , M.D. (Individual)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Gary M Levine, M.D., Director of Breast Imaging, Levine, Gary M. , M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-01-LEV
Record Dates: First submitted 2011-06-02; First posted 2011-06-23 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Radiography; Breast Specimen Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast biopsy specimen imaging & comparison of image quality (Experimental): Each subject's explanted tissue will serve as both the control (standard analysis) and the experimental analysis of the quality of the images.
  Interventions: Device: Trident Specimen Radiography System; Device: Bioptics, Faxitron, and Full Field Digital Mammography (FFDM) Selenia

INTERVENTIONS:
Device: Trident Specimen Radiography System — MIBB images will be acquired on the standard of care device and the Trident System in the Breast Center at Hoag Hospital. BSS images will be acquired on standard of care device in the Operating Room and/or the Breast Center at Hoag Hospital and then on the Trident System. Image quality will be compared and system operation will be evaluated. Feedback will be provided to manufacturer and the Trident System further refined.
Device: Bioptics, Faxitron, and Full Field Digital Mammography (FFDM) Selenia — All the above devices are used for SOC BSS imaging at Hoag Hospital. The images captured from these devices will be compared to the images captured from the Trident Specimen Radiography device.

SUMMARY:
The objective of this study is to evaluate the image quality and operation of a self-contained direct digital radiography system for breast specimen imaging.

DETAILED DESCRIPTION:
Specimen imaging is an accepted method for evaluating tissue specimens which are obtained either through minimally-invasive breast needle biopsy (MIBB) or breast surgery. Specimen imaging is used to confirm the targeting and sampling adequacy of radiographically apparent breast abnormalities. Specimen images are acquired and then compared to the routine and diagnostic imaging to provide radiographic evidence that the index lesion was adequately targeted and sampled (as in the case of MIBB) or targeted and removed with adequate margins [as in the case of breast surgical specimens (BSS)]. Specimen imaging also provides guidance to the histopathologist when evaluating the breast specimen.

Near real-time image acquisition, review and feedback is essential for specimen imaging. The patient typically remains in compression on the biopsy table for MIBB or under anesthesia for BSS until the clinician has confirmation that the index abnormality has been adequately sampled (in the case of MIBB) or surgically excised. For this reason, digital techniques are favored over analog (film) counterparts because of the immediacy of image acquisition and transfer and display to the radiologist for review.

Image quality and speed are critical factors in specimen imaging. High resolution images are a clinical requirement to delineate the features and extent of mass lesions, and presence and extent of microcalcifications.

Conventional full-field digital (FFDM) mammographic equipment located in the mammography department is one accepted approach for specimen imaging. An advantage of this method is that a licensed and skilled mammographic technologist assures the adequate exposure of specimens. However, this method requires that the FFDM system be free at the time the specimen arrives in the mammography department, interfering with mammogram schedules. In the case of BSS, the use of conventional FFDM systems additionally requires the transport of specimens to the mammography department, adding significant time that the patient is under anesthesia.

Another mode for specimen radiography is self-contained digital radiography specimen imaging systems that are located in the mammography department or in the Operating Room (intraoperative). The use of self-contained digital systems frees the conventional mammography system for its intended purpose, while providing the clinician all the speed of digital radiography.

It has been shown that intraoperative imaging significantly reduces the amount of time that the patient is under anesthesia.

Although, self-contained digital radiography specimen imaging systems provide an advantage in speed, resulting images may suffer in image quality and despite the availability of intraoperative self contained systems, many clinicians choose to transfer specimens to the mammography department for imaging on a conventional FFDM system. Current specimen radiography systems employ an indirect digital technique, a two step conversion, where incoming x-ray signal is converted to light and then to digital signal. The intermediate step of converting signal to light, leads to diffusion and scatter over many pixels and this in turn leads to degradation of the very fine features of mass densities and microcalcifications.

Direct Digital technique is another method currently used in breast imaging. The direct digital technique has the advantage of converting incoming signal directly to digital signal, avoiding the intermediary light conversion phase of indirect exposure. The direct to digital process results in better use of incoming signal and greater resolution and thus a sharper image, providing high resolution of minute features associated with mass lesions and microcalcifications.

Another common characteristic of current self-contained systems is the use of "stitching" many small CMOS chips to create a larger image detector. This type of tiling provides for a more economical system, but shearing effects, gaps between chips and overall concerns with calibration of multiple chips significantly degrades image quality.

All digital images, indirect or direct are acquired in a raw state and processed to allow review. While image processing cannot improve or change the raw aspects of the image after acquisition, processing can improve the visibility of features available in the image. Image processing is fundamentally associated with image acquisition technique. If the image is not adequately exposed, image processing will not be optimally applied and in some cases fail, requiring additional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Breast specimens acquired through MIBB or Surgical techniques arriving for specimen imaging

Exclusion Criteria:

* Breast specimens that are larger than12 x 14 cm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Breast biopsy specimen will be imaged on standard of care device and on the Trident Specimen Radiography device to compare quality of images. | 1 Day
  Images will be taken at time of biopsy with no additional follow-up time for patient.

SECONDARY OUTCOMES:
Device Operation | 1 Day
  Device will be evaluated for length of time to carry out procedure, ease of use in patient data entry, procedure selection, taking the exposure, usability and usefulness of image manipulation tools and overall rating.

CONTACTS AND LOCATIONS:
Overall Officials: Gary M. Levine, M.D., Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Background] Silverstein MJ, Lagios MD, Recht A, Allred DC, Harms SE, Holland R, Holmes DR, Hughes LL, Jackman RJ, Julian TB, Kuerer HM, Mabry HC, McCready DR, McMasters KM, Page DL, Parker SH, Pass HA, Pegram M, Rubin E, Stavros AT, Tripathy D, Vicini F, Whitworth PW. Image-detected breast cancer: state of the art diagnosis and treatment. J Am Coll Surg. 2005 Oct;201(4):586-97. doi: 10.1016/j.jamcollsurg.2005.05.032. No abstract available. PMID 16183499
- [Background] Kaufman CS, Jacobson L, Bachman BA, Kaufman LB, Mahon C, Gambrell LJ, Seymour R, Briscoe J, Aulisio K, Cunningham A, Opstad F, Schnell N, Robertson J, Oliver L. Intraoperative digital specimen mammography: rapid, accurate results expedite surgery. Ann Surg Oncol. 2007 Apr;14(4):1478-85. doi: 10.1245/s10434-006-9126-5. Epub 2007 Jan 18. PMID 17235716